CLINICAL TRIAL: NCT03624686
Title: Production of Clinical-grade Anti-CD19 Chimeric Antigen Receptor T Cells for Refractory B-cell Malignancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201711021RIND
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-03

CONDITIONS: Leukemia
Keywords: Acute Lymphoblastic Leukemia,Immunotherapy,chimeric antigen receptor,non-Hodgkin's lymphoma
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy volunteer
  Interventions: Other: peripheral blood
- luekemia patient
  Interventions: Other: peripheral blood

INTERVENTIONS:
Other: peripheral blood — draw peripheral blood

SUMMARY:
Immunotherapy is a promising therapeutic approach for patients with cancers. Patients with acute lymphoblastic leukemia (ALL) experiencing early relapse less than 18 months from diagnosis had very poor prognosis with 5-year survival rate of 21% (1). Recent clinical trials demonstrated that infusions of autologous T cell modified with chimeric antigen receptors (CARs) induced durable complete remissions in patients with relapse or refractory B-cell ALL (2-4). The editors of Science Journal announced cancer immunotherapy as the breakthrough of the year for 2013 (5). On Jan 30, 2015, Dr. Steven M. Altschuler, chief executive officer of the Children's Hospital of Philadelphia and 9-year-old ALL patient Emily Whitehead with 3-year leukemia free after CAR-T cell infusion were invited to White House for President Barack Obama's announcement of the Precision Medicine Initiative. The MIT Technology Review announced that the top one breakthrough technology in 2016 is genetically engineered immune cells saving the lives of cancer patients. This project will focus on the manufacturing of clinical-grade anti-CD19 CARs for B-cell malignancies in the future clinical trials.

ELIGIBILITY:
1. At least 14 years of age (underage patients under the age of 20 only collect peripheral venous blood, do not perform double-lumen venous catheter and white blood cell separation).
2. There are no known serious systems or diseases with systemic immunodeficiency, but blood-related cancers are not.
3. Systemic chemotherapy and target treatment were not received within 14 days.
4. The subject consent form has been signed prior to the program-related procedures.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Leukemia patients and healthy volunteer aged 14 and over
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-03-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Clinical process of CAR-T cells | JAN/2018-DEC/2020
  Establish a clinical process for CAR-T cells in the GTP laboratory and document these steps to establish a complete standard operation procedure (SOP) and further validate the process to comply with GMP regulations

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Chang, MDPHD, Principal Investigator — natinal taiwan university hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan